CLINICAL TRIAL: NCT01613664
Title: Randomized Prospective Clinical Study Evaluating the Usefulness of Fibrin Glue (TISSEEL® KIT) to Prevent Gastric Fistula, Intra Abdominal Haemorrhage and Intra Abdominal Loco Regional Collections After Laparoscopic Sleeve Gastrectomy
Brief Title: Efficiency of TISSEEL for Sleeve Gastrectomy Complications
Acronym: TISSEEL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI11-PR-REGIMBEAU-2
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Morbid Obesity
Keywords: obesity; surgical management; sleeve gastrectomy
MeSH Terms: conditions — Obesity, Morbid; Obesity | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tisseel (Experimental): tisseel will be applied during the surgery
  Interventions: Drug: tisseel
- no tisseel (Placebo Comparator): no tisseel will be applied during the surgery
  Interventions: Other: no tisseel

INTERVENTIONS:
Drug: tisseel — The product will be given as a 2 mL bottle per patient, which will be spread along the staple line. If necessary, a second bottle of 2 mL is used. The precautions for use are described in the user manual.
  Arms: tisseel
Other: no tisseel — the surgeon does not applied tissucol during the surgery
  Arms: no tisseel

SUMMARY:
Laparoscopic Sleeve Gastrectomy has emerged over the last 20 years as a treatment of choice in the surgical management of patients with morbid obesity. However, this restrictive procedure is accompanied by outcomes such as gastric fistula (5%), postoperative hemorrhage (1%) and intra-abdominal loco regional collections (1%). At present, there is no sufficiently reliable technique to prevent these complications.

DETAILED DESCRIPTION:
The hypothesis is the following : the use of fibrin glue (Tissucol ®) during Laparoscopic Sleeve Gastrectomy would reduce the incidence of complications (gastric fistula, intra-abdominal hemorrhage and intra-abdominal locoregional collection).

The aim is to investigate whether the use of fibrin glue (Tissucol®) during Laparoscopic Sleeve Gastrectomy reduces the incidence of postoperative complications (gastric fistula, intra-abdominal hemorrhage and intra-abdominal locoregional collection)

ELIGIBILITY:
Inclusion Criteria:

* Obesity requiring bariatric surgery (Laparoscopic Sleeve Gastrectomy) according to the Haute Autorité de Santé
* Patients younger than 60 years old
* BMI ≤ 60 kg/m2
* Surgery accepted by an Obesity-related specific committee
* Patient with social protection

Exclusion Criteria:

* Previous bariatric or gastric surgery
* BMI > 60 kg/m2
* Under 18 years old
* Allergy to Tissucol®
* peroperative fistula
* Consent not signed
* Incapable of giving his opinion
* Pregnancy or breast-feeding
* Contraindication to surgery
* ASA classification IV

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 597 (Actual)
Dates: Start 2014-02; Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
presence of post-operative complications | post operative day 30
  The primary endpoint corresponds to the presence of complications after laparoscopic sleeve gastrectomy during the follow up period. A complication is considered as "present" if at least one of the following three items is present:
  * Gastric fistula
  * Postoperative hemorrhage
  * intra-abdominal locoregional collection

SECONDARY OUTCOMES:
The gastric fistula's rate | post operative day 30
The postoperative hemorrhage's rate | post-operative day 30
The intra-abdominal locoregional collection's rate | post-operative day 30
the length of stay | post-operative day 30
the rate of readmission | post-operative day 30
the rate of reintervention | post-operative day 30
the overall mortality at one month | post-operative day 30
the specific mortality at one month | post-operative day 30
the rate of postoperative morbidity | postoperative day 30
  the morbidity will be evaluated according to the clavien dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc REGIMBEAU, MD,phD, Principal Investigator — chu amiens; michel scotte, MD PhD, Principal Investigator — chu Rouen
Locations (2):
- France (2):
  - North Universitary Hospital, Amiens
  - Charles Nicolle Universitary Hospital, Rouen

REFERENCES:
- [Background] Pequignot A, Fuks D, Verhaeghe P, Dhahri A, Brehant O, Bartoli E, Delcenserie R, Yzet T, Regimbeau JM. Is there a place for pigtail drains in the management of gastric leaks after laparoscopic sleeve gastrectomy? Obes Surg. 2012 May;22(5):712-20. doi: 10.1007/s11695-012-0597-0. PMID 22328096
- [Background] Pequignot A, Dhahria A, Mensah E, Verhaeghe P, Badaoui R, Sabbagh C, Regimbeau JM. Stapling and Section of the Nasogastric Tube during Sleeve Gastrectomy: How to Prevent and Recover? Case Rep Gastroenterol. 2011;5(2):350-4. doi: 10.1159/000329706. Epub 2011 Jul 6. PMID 21769286
- [Background] Dhahri A, Verhaeghe P, Hajji H, Fuks D, Badaoui R, Deguines JB, Regimbeau JM. Sleeve gastrectomy: technique and results. J Visc Surg. 2010 Oct;147(5 Suppl):e39-46. doi: 10.1016/j.jviscsurg.2010.08.016. No abstract available. PMID 20971049
- [Background] Sabbagh C, Verhaeghe P, Dhahri A, Brehant O, Fuks D, Badaoui R, Regimbeau JM. Two-year results on morbidity, weight loss and quality of life of sleeve gastrectomy as first procedure, sleeve gastrectomy after failure of gastric banding and gastric banding. Obes Surg. 2010 Jun;20(6):679-84. doi: 10.1007/s11695-009-0007-4. Epub 2009 Nov 10. PMID 19902316
- [Background] Fuks D, Verhaeghe P, Brehant O, Sabbagh C, Dumont F, Riboulot M, Delcenserie R, Regimbeau JM. Results of laparoscopic sleeve gastrectomy: a prospective study in 135 patients with morbid obesity. Surgery. 2009 Jan;145(1):106-13. doi: 10.1016/j.surg.2008.07.013. Epub 2008 Sep 30. PMID 19081482
- [Derived] Rebibo L, Dhahri A, Chati R, Cosse C, Huet E, Regimbeau JM. Effectiveness of Fibrin Sealant Application on the Development of Staple Line Complications After Sleeve Gastrectomy: A Prospective Randomized Trial. Ann Surg. 2018 Nov;268(5):762-768. doi: 10.1097/SLA.0000000000002892. PMID 30080735